CLINICAL TRIAL: NCT06943131
Title: Comparison of YWTL Exercises and Closed Kinetic Chain Exercises on Shoulder Pain, Disability, Upper Limb Mobility and Posture in Children With Scapular Dyskinesis.
Brief Title: YWTL Exercises and Close Kinetic Chain Exercises in Children With Scapular Dyskinesis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/24/0728
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Scapular Dyskinesis
Keywords: Scapular Dyskinesis, Scapulohumeral YWTL Exercises.

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial will be performed, in which 22 children with scapular dyskinesis with age 9 to 12 years will be taken after screening and meeting inclusion criteria. children will be divided into 2 groups. group 1 will receive YWTL exercises for alternating 3 days a week. Group 2 will receive closed kinetic chain exercises for alternating 3 days a week. Pre values were taken at 1st week and then post values of intervention will be taken after 6th week of intervention to measure the effect of both therapies.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 with YWTL exercises (Experimental): group 1 will receive YWTL exercises for alternating 3 days a week for 6 weeks.
  Interventions: Other: YWTL EXERCISES; Other: Closed kinetic chain exercises
- group 2 with closed kinetic chain exercises (Experimental): group 2 will receive closed kinetic chain exercises for alternating 3 days a week for 6 weeks.
  Interventions: Other: YWTL EXERCISES; Other: Closed kinetic chain exercises

INTERVENTIONS:
Other: YWTL EXERCISES — YWTL exercises are shoulder and upper back exercises to improve posture, strengthen upper back. Each letter represents different arm position that copies shape of letter.
Other: Closed kinetic chain exercises — Closed kinetic chain exercises include corner stretch hold, sleeper stretch hold - lawn mover and robbery maneuver, Scapula clock exercises, wall wash. Low row exercise maneuver, Scapular stabilization of Black burn exercises, press up, push up.

SUMMARY:
Scapular dyskinesia is defined by abnormal movement or placement of the scapula, the shoulder blade, during arm movements. Physical treatment aimed at regaining appropriate scapular mechanics through strengthening exercises, postural correction, and functional movement training is typically part of management. A randomized clinical trial will be conducted. The study will be conducted at Unique school and on school going children in a total duration of 10 months. Sample size will be 22.There will be two study groups. A convenient sampling technique will be used. The sample which will have following characteristics will be included children with age group 9 to 12 years, positive scapular test, positive scapular assistance test, athletes who practice one hour three days a week. The sample with the following characteristics will be excluded. Any muscular or joint deformity, scoliosis, shoulder dislocation. The tools that will be included in the study are modified lateral scapular test, shoulder flexion test, shoulder and pain disability index, upper extremity functional use scale, posture and posture assessment scale, shoulder and scapular ranges.

DETAILED DESCRIPTION:
Scapular dyskinesia is defined by abnormal movement or placement of the scapula, the shoulder blade, during arm movements. Changes in scapular kinematics, such as tipping (forward or backward tilting), winging (medial border protrusion), or general prominence during shoulder movements, are usually involved. Physical treatment aimed at regaining appropriate scapular mechanics through strengthening exercises, postural correction, and functional movement training is typically part of management. From the shoulders to the hands, proper upper limb posture is essential for both biomechanical effectiveness and the avoidance of injuries when performing tasks. In addition to maximizing mobility for daily tasks, work, sports, and leisure activities, proper posture relieves tension on muscles and joints, assuring effective performance and lowering the chance of injury. A randomized clinical trial will be conducted. The study will be conducted at Unique School Wapda Town and The Punjab School in a total duration of 10 months. Sample size will be 22.

There will be two study groups. A convenient sampling technique will be used. The sample which will have following characteristics will be included children with age group 9 to 12 years, positive scapular test, positive scapular assistance test, normal shoulder ranges, normal scapular ranges, athletes who practice one hour three days a week. The sample with the following characteristics will be excluded. Any muscular or joint deformity, scoliosis, shoulder dislocation, previous surgery of shoulder and cervicobrachialgia. The tools that will be included in the study are modified lateral scapular test, scapular dyskinesis test, shoulder flexion test, scapular assistance test, shoulder and pain disability index, upper extremity functional use scale, posture and posture assessment scale, shoulder and scapular ranges. SPSS version 27 will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

Children with an age group of 9 to 12 years.

* Both genders.
* Engage in overhead sports.
* Minimum play time is 1 hour 3 times in a week.
* Positive Modified lateral scapular test
* Positive scapular dyskinesis shoulder flexion test
* Positive scapular assistance test
* Shoulder and pain disabilty index (score 1 to 20 )
* Upper extremity functional use scale (score 60 to 80).

Exclusion Criteria:

Any muscular or joint deformity.

* Scoliosis.
* Shoulder dislocation
* Post fracture.
* Neurological deficits
* Cervicobrachialgia

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
modified lateral scapular test | pre reading(1st week) post reading (6th week)
  The Modified Lateral Scapular Slide Test assesses scapular asymmetry and stability by measuring the distance between the inferior angle of the scapula and the spine in various arm positions.
scapular dyskinesis test | pre reading(1st week) post reading (6th week)
  The Scapular Dyskinesis Test evaluates abnormal scapular movement patterns during shoulder motion to identify dysfunction.
shoulder flexion test | pre reading(1st week) post reading (6th week)
  The Shoulder Flexion Test assesses the range of motion and flexibility of the shoulder joint as the arm is raised overhead.
scapular assistance test | pre reading(1st week) post reading (6th week)
  The Scapular Assistance Test evaluates the effect of manually assisting scapular motion on shoulder pain and function during arm elevation.
shoulder and pain disability index | pre reading(1st week) post reading (6th week)
  The Shoulder Pain and Disability Index (SPADI) is a self-reported questionnaire that measures the pain and functional impairment associated with shoulder disorders.
upper extremity functional use scale | pre reading(1st week) post reading (6th week)
  The Upper Extremity Functional Use Scale assesses the frequency and quality of functional use of the affected upper limb in daily activities.
posture and posture assessment scale | pre reading(1st week) , post reading (6th week)
  The Posture and Postural Ability Scale includes items for measuring posture as well as a 7-point ordinal scale for postural ability in supine, prone, sitting, and standing
shoulder ranges | pre reading(1st week) , post reading (6th week)
  Shoulder ranges refer to the degrees of motion the shoulder joint can achieve in various directions, including flexion, extension, abduction, adduction, and rotation.
scapular ranges | pre reading(1st week), post reading (6th week)
  Scapular ranges are the measurable degrees of movement the scapula performs during shoulder motions, including elevation, depression, protraction, retraction, and rotation.

CONTACTS AND LOCATIONS:
Overall Officials: Mishal Farwa, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Mishal Farwa, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teixeira DC, Alves L, Gutierres M. The role of scapular dyskinesis on rotator cuff tears: a narrative review of the current knowledge. EFORT Open Rev. 2021 Oct 19;6(10):932-940. doi: 10.1302/2058-5241.6.210043. eCollection 2021 Oct. PMID 34760292
- [Background] Hogan C, Corbett JA, Ashton S, Perraton L, Frame R, Dakic J. Scapular Dyskinesis Is Not an Isolated Risk Factor for Shoulder Injury in Athletes: A Systematic Review and Meta-analysis. Am J Sports Med. 2021 Aug;49(10):2843-2853. doi: 10.1177/0363546520968508. Epub 2020 Nov 19. PMID 33211975
- [Background] Otoshi K, Kikuchi S, Kato K, Sato R, Igari T, Kaga T, Konno S. The prevalence of scapular malalignment in elementally school aged baseball player and its association to shoulder disorder. J Orthop Sci. 2018 Nov;23(6):942-947. doi: 10.1016/j.jos.2018.07.006. Epub 2018 Aug 4. PMID 30087015
- [Background] 4. Mahale A, Bisen R, Kalra K. Prevalence of Scapular Dyskinesia in Elite Badminton Players in Pune. International Journal of Health Sciences and Research. 2020;10(11):127-34.
- [Background] Joseph R, Alenabi T, Lulic T, Dickerson CR. Activation of Supraspinatus and Infraspinatus Partitions and Periscapular Musculature During Rehabilitative Elastic Resistance Exercises. Am J Phys Med Rehabil. 2019 May;98(5):407-415. doi: 10.1097/PHM.0000000000001116. PMID 30550457
- [Background] Gianakos AL, Abdelmoneim A, Kerkhoffs G, Mulcahey MK. Rehabilitation and Return to Sport of Female Athletes. Arthrosc Sports Med Rehabil. 2022 Jan 28;4(1):e247-e253. doi: 10.1016/j.asmr.2021.09.040. eCollection 2022 Jan. PMID 35141558